CLINICAL TRIAL: NCT01043770
Title: A Randomised Controlled Trial to Investigate the Effects of a Structured Self-management Education Programme for People With Metabolic Syndrome
Brief Title: The Reversal Intervention for Metabolic Syndrome Study
Acronym: TRIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0025
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2011-12

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Primary prevention; Diabetes; Cardiovascular disease; Patient education
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group lifestyle education (Experimental): Multi-component behaviour change intervention
  Interventions: Behavioral: Group lifestyle education
- Routine care (No Intervention): Routine care

INTERVENTIONS:
Behavioral: Group lifestyle education — Structured group education programme based on lifestyle changes (dietary and increased physical activity)
  Arms: Group lifestyle education

SUMMARY:
The aim of our study is to see if people with metabolic syndrome who attend a group education programme based on lifestyle changes (dietary and increased physical activity) can lessen their risk of having diabetes, heart disease and strokes in the future.

DETAILED DESCRIPTION:
People who have a combination of risk factors termed metabolic syndrome are at increased risk of developing diabetes, heart disease and strokes. Metabolic syndrome is a major public health concern requiring urgent action because 25% of the adult UK population fulfil the criteria, and this will increase as people continue to be less active and levels of overweight and obesity rise.

The aim of our study is to see if people with metabolic syndrome who attend a structured group education programme based on lifestyle changes (dietary and increased physical activity) can lessen their risk of having diabetes and cardiovascular disease in the future. Overall, we hope to show that this type of education reduces the number of people who have metabolic syndrome.

Subjects recruited with metabolic syndrome will be randomised to intervention or control arms. The intervention arm will receive group education and the control group will receive routine care.

The results will inform primary prevention strategies in people from varied ethnic backgrounds who are at high risk of developing type-2 diabetes and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 - 74 years inclusive
* Registered with a general practice in Leicester City or Leicester County Primary Care Trust
* Availability of data to allow diagnosis of MetS (IDF criteria) collected at a screening visit

Exclusion Criteria:

* Previous diagnosis of T2DM, CVD (stroke/cerebrovascular accident, transient ischaemic attack), peripheral arterial disease, or coronary heart disease (angina, myocardial infarction, coronary artery bypass surgery, angioplasty)
* Life-limiting terminal illness
* Pregnancy and/or breast feeding
* Lack of capacity to give informed consent because of serious mental health problems or learning disability.
* People who are housebound
* Patients residing in nursing/care homes
* Individuals who are unable to speak and understand English. (The intervention will be made appropriate for ethnically diverse populations, but individuals who are unable to understand, speak and read English will be excluded at this stage. However, if the self-management programme is found to be successful we would adapt it for non-English speakers.)

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The proportion of people in the intervention and control groups with prevalent metabolic syndrome according to the IDF criteria. | 12 months follow-up.

SECONDARY OUTCOMES:
The prevalence of metabolic syndrome according to NCEP criteria | Compared at baseline versus 12 months, and for the intervention group versus the control group
Changes in individual components of the metabolic syndrome (fasting plasma glucose, triglycerides, HDL cholesterol, blood pressure, waist circumference), and 2 hour glucose | Compared at baseline versus 12 months, and for the intervention group versus the control group
Changes in biomarkers (hs-CRP, adiponectin, and insulin) | Compared at baseline versus 12 months, and for the intervention group versus the control group
Changes in physical activity as measured by IPAQ and pedometer | Compared at baseline versus 12 months, and for the intervention group versus the control group
Changes in dietary/nutritional intake measured by DINE | Compared at baseline versus 12 months, and for the intervention group versus the control group
Changes in Framingham risk score | Compared at baseline versus 12 months, and for the intervention group versus the control group
Changes in quality of life as measured by EuroQol EQ-5D | Compared at baseline versus 12 months, and for the intervention group versus the control group
Changes in depression/anxiety as measured by HADS | Compared at baseline versus 12 months, and for the intervention group versus the control group
Changes in general self-efficacy as measured by GSE | Compared at baseline versus 12 months, and for the intervention group versus the control group

CONTACTS AND LOCATIONS:
Overall Officials: Kamlesh Khunti, MD, FRCGP, Principal Investigator — Diabetes Research Centre, University of Leicester; Melanie J Davies, MD, FRCP, Principal Investigator — Diabetes Research Centre, University of Leicester
Locations (1):
- University of Leicester, Leicester, United Kingdom

REFERENCES:
- [Result] Dunkley AJ, Davies MJ, Stone MA, Taub NA, Troughton J, Yates T, Khunti K. The Reversal Intervention for Metabolic Syndrome (TRIMS) study: rationale, design, and baseline data. Trials. 2011 May 4;12:107. doi: 10.1186/1745-6215-12-107. PMID 21542913